CLINICAL TRIAL: NCT06899919
Title: Evaluation of the Efficacy and Safety of Light Compression System Versus Tubular Bandage in the Local Treatment of Mixed Leg Ulcers: a Prospective Open-label RCT
Brief Title: Efficacy and Safety of Light Compression System in the Local Treatment of Mixed Leg Ulcers (PROMETHEE Clinical Investigation)
Acronym: PROMETHEE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoires URGO (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID RBC : 2024-A01402-45
Record Dates: First submitted 2025-03-21; First posted 2025-03-28 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Leg Ulcers
Keywords: Mixed leg ulcers; Quality of life questionnaire; light compression system
MeSH Terms: conditions — Leg Ulcer | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: randomization 2:1 (light compression system vs tubular bandage)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- light compression system (Experimental): Treatment with two bandages light compression system during 16-week treatment period (6 medical visits are planned: D0, W2, W4, W8, W12, W16)
  Interventions: Device: Treatment with light compression systeme during 16-week treatment period (6 medical visits are planned: D0, W2, W4, W8, W12, W16); Device: Light compression system of the mixed leg ulcer stage C6 / C6r of the CEAP classification
- tubular bandage (Placebo Comparator): Treatment with tubular bandage system during 16-week treament period (6 medical visits are planned: D0, W2, W4, W8, W12, W16)
  Interventions: Device: Treatment with light compression systeme during 16-week treatment period (6 medical visits are planned: D0, W2, W4, W8, W12, W16); Device: Light compression system of the mixed leg ulcer stage C6 / C6r of the CEAP classification

INTERVENTIONS:
Device: Treatment with light compression systeme during 16-week treatment period (6 medical visits are planned: D0, W2, W4, W8, W12, W16) — Treatment with light compression system during 16-week treatment period (6 medical visits are planned: D0, W2, W4, W8, W12, W16)
Device: Light compression system of the mixed leg ulcer stage C6 / C6r of the CEAP classification — Etiological treatment of mixed leg ulcer stage C6 / C6r of the CEAP classification

SUMMARY:
Evaluation of the efficacy (wound epithelialization and time to closure) and safety (emergence and nature of adverse event) of a lite compression system versus a tubular bandage in the local treatment of mixed leg ulcers: prospective multicenter, randomized controlled, open-label french clinical study

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled, open-label, multicenter clinical trial conducted in patients with a mixed (non-ischemic) leg ulcer of stage C6 / C6r of the CEAP classification.

This study is carried out in around 50 French investigational centers. A total of 210 patients meeting the eligibility criteria will be included. The patients will be followed for 16 weeks and a total of 6 clinical evaluations will be carried out by the investigating centers.

A planimetric survey of the studied leg ulcers is carried out during the initial assessment of the wound (Day 0) and at each assessment provided for in the protocol (Week 2, Week 4, Week 8 and Week 12).

A QoL is carried out at D0 and end of the study for each patient included in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥ 18 years old), having given free, informed and written consent
* Patient affiliated to a social security scheme
* Patient agreeing to wear the study compression system daily
* Patient with an ankle circumference between 18 and 25 cm
* Target wound: stage C6 / C6r mixed leg ulcer of the CEAP classification with a 0.6≤ ABPI≤0.8 and TABP≥ 50 mm Hg and arterial echo Doppler confirming the mixed nature of the leg ulcer
* Target wound with an area between 2 and 20 cm2
* Target wound with age of ≤18 months

Criteria exclusion:

* Patient with a systemic infection not controlled by appropriate antibiotic therapy
* Patient having presented in the 3 months preceding his inclusion, a deep vein thrombosis
* Severe arterial pathology, including an Ankle Blood Pressure Index (ABPI) less than 3 months old <0.6
* Patient bedridden or spending less than an hour per day standing
* Clinically infected target wound
* Cancerized target wound

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-03-29 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Complete closure of the Venous Leg Ulcer (VLU) | 16-week treament period
  Description: Complete closure of the leg ulcer is defined by 100% re-epithelialization of the mixed Leg Ulcer (MLU)

SECONDARY OUTCOMES:
Time to complete closure of the Venous Leg Ulcer (VLU) | 16-week treament period
  Description: Time to complete closure of the Mixed Leg Ulcer (MLU) is defined as the time from inclusion to the date of complete closure
Safety analysis | 16-week treament period
  Nature and number of adverse event related to the use of the studied light compression system and tubular bandage (serious/ non-serious and emergent)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia PaS SENET, Dr, MD, PhD, Principal Investigator — Hôpitaux Universitaires Paris Est (AP-HP) - Hôpital TENON
Locations (3):
- France (3):
  - Patricia SENET, Paris, Paris 75000, Paris, Paris
  - Cabinet d'Angiologie - Médecine Vasculaire 377 rue Garibaldi 69007 LYON, Lyon
  - APHP Hopital TENON Service de Dermatologie et médecine vasculaire 4 Rue de la Chine 75970 PARIS Cedex 20, Paris